CLINICAL TRIAL: NCT05902793
Title: Prospective, Multi-center, Randomized, Open Label, Parallel Group Controlled, Non-inferiority Trial Evaluating the Efficacy and Safety of the VERAFLO™ Dressing Kit for Wound Bed Preparation in Open Wounds With Extensive Soft Tissue Damage
Brief Title: Evaluating the Efficacy and Safety of the VERAFLO™ Dressing Kit for Wound Bed Preparation in Open Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KCI USA, Inc (Industry)
Responsible Party: Sponsor
Organization: Solventum US LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EM-05-015052
Record Dates: First submitted 2023-05-01; First posted 2023-06-15 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Wound Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Investigational device: V.A.C. VERAFLO™ Dressing Kit (Experimental): NPWT consists in applying topical sub-atmospheric pressure to a wound that is covered with V.A.C. VERAFLO™ Dressing, sealed with drape and connected by a tube to a suction pump applying -125mmhg pressure with a drainage collection system. Instillation and dwell of a topical wound solution in the wound bed cycled at set intervals of 10 minutes every 3.5 hours without negative pressure applied. The target wound for each subject in both groups will be treated for up to 14 days or until deemed ready for closure by the investigator (whichever occurs first).
  Interventions: Device: Investigational device: V.A.C. VERAFLO™ Dressing Kit
- Negative pressure wound drainage material (Active Comparator): A Negative pressure wound drainage material manufactured by Guangdong Shuangling Pharmaceutical Co., Ltd. (with unspecified pressures ranging from -150 to -380mmHg ) was selected as the control group treatment device, which can apply the NPWT therapy with wall suction. This control device is widely used in clinical institutions in China to deliver NPWT. The target wound for each subject in both groups will be treated for up to 14 days or until deemed ready for closure by the investigator (whichever occurs first).
  Interventions: Device: Comparator device: Negative pressure wound drainage material

INTERVENTIONS:
Device: Investigational device: V.A.C. VERAFLO™ Dressing Kit — Up to 170 subjects who meet the eligibility criteria will be randomized to the investigational group or control group at the ratio 1:1.
  Subjects will only be enrolled following definitive surgical debridement (if serial debridement performed) of the target wound. The target wound for each subject in both groups will be treated for up to 14 days or until deemed ready for closure by the investigator (whichever occurs first). The planned study period consists of the following visits: Screening (Day -3 to 0), Day of randomization (Day0), Dressing change visit(s), End of treatment visit. Following study treatment, the wound may be treated with any standard therapy selected by the physician, and then accepted secondary intervention for wound closure according to the wound bed preparation situation.
  Arms: Investigational device: V.A.C. VERAFLO™ Dressing Kit
Device: Comparator device: Negative pressure wound drainage material — Up to 170 subjects who meet the eligibility criteria will be randomized to the investigational group or control group at the ratio 1:1.
  Subjects will only be enrolled following definitive surgical debridement (if serial debridement performed) of the target wound. The target wound for each subject in both groups will be treated for up to 14 days or until deemed ready for closure by the investigator (whichever occurs first). The planned study period consists of the following visits: Screening (Day -3 to 0), Day of randomization (Day0), Dressing change visit(s), End of treatment visit. Following study treatment, the wound may be treated with any standard therapy selected by the physician, and then accepted secondary intervention for wound closure according to the wound bed preparation situation.
  Arms: Negative pressure wound drainage material

SUMMARY:
The objectives are to evaluate the efficacy and safety of the V.A.C. VERAFLO™ Dressing Kit for wound bed preparation in open wounds with extensive soft tissue damage in this trial.

DETAILED DESCRIPTION:
The management of wounds represents a significant challenge in healthcare. There are many considerations necessary in developing the optimal treatment plan for achieving wound care goals. Current standard wound treatment in the management of wounds may involve clinical assessment, debridement, antibiotic treatment and local application of antiseptics or antimicrobials, and drainage.

The choice of therapeutic modality is one of many important decisions. Over time, wound care has progressed from the use of products such as dry gauze to advanced moist wound therapies and further to active wound healing therapies. One of such advanced wound healing therapies is negative pressure wound therapy (NPWT), which was developed in the 1990s. NPWT is a technology that is currently widely used in wound care and is promoted for use on complex wounds (open wounds). The therapy of NPWT and solution instillation with a dwell time (NPWTi-d) is used to adjunctively treat high-risk wounds that would benefit from vacuum-assisted drainage and controlled repeated delivery of topical wound solutions, such as normal saline and wound cleansers. Evidences suggests that normal saline is effective and readily available.

V.A.C. VERAFLO™ Dressing Kit, which was the investigational device, was a reticulated open-cell foam polyurethane ester dressing that could deliver normal saline instillation solution to the wound site for NPWTi-d therapy. The V.A.C. VERALFO™ Dressing Kit was approved in July 2010 by the U.S Food and Drug Administration (U.S. FDA) and December 2022 by the China National Medical Products Administration (NMPA).

This trial was designed as a pre-marketing trial of the V.A.C. VERAFLO™ Dressing Kit in China for NMPA registration. The device V.A.C. VERALFO™ Dressing Kit did not get NMPA approval when the study was initiated. On December 20th, 2022, it was approved by NMPA (Registration No.: 国械注进 20223140619).

There were no approved NPWTi-d dressings in China market during protocol design, so a negative pressure wound drainage material manufactured by Guangdong Shuangling Pharmaceutical Co., Ltd. was selected as the control group treatment device, which can apply the NPWT therapy with wall suction.

ELIGIBILITY:
Inclusion Criteria:

Only adult subjects meeting all of the following criteria to be considered for participation:

1. Subject voluntarily participate in the trial and sign the informed consent form, and is willing to comply with protocol and all visits
2. Is anticipated to be an inpatient for a minimum of 6 days
3. Age: between 18 years and 70 years
4. Patient with open wounds from various etiologies with extensive soft tissue damage after definitive surgical debridement and appropriate for NPWT
5. The minimum size of the wound as measured by 3D wound imaging prior to entry into the study is 8cm (in any dimension), minimum 1cm in width and 0.8cm in depth. i.e. the minimum wound size is 8cm×1cm×0.8cm. Only one wound per subject will be included in the study, regardless of how many wounds the subject has.
6. Female subjects of reproductive potential must have a negative pregnancy test result and must not be lactating at the screening visit.
7. Subject must be willing and able to use a highly effective contraception method during study participation.

Exclusion Criteria:

Subject who meets any of the following criteria will be excluded from participation in the study:

1. Subject undergoing chemotherapy
2. Subject with known immunodeficiency
3. Subject with serious complications or serious systemic infection
4. Known bleeding disorder or has received or is planning to receive long-term anticoagulation therapy
5. Known allergic reactions/hypersensitivity to any of the study treatment dressings components
6. Target wound is a burn wound
7. A wound open for 6 months or more
8. The subject's targeted traumatic wound injury is a craniofacial wound
9. There is implant (such as cardiac pacemaker, bone nail, bone lamella, artificial joint, artificial bone) visible in the targeted wound.
10. If undermining or tunneling represents approximately 15% or more of the wound.
11. A wound with enteric fistulas.
12. Subject's targeted wound that is contraindicated with investigational device including:

    1. Malignancy in the wound
    2. Untreated osteomyelitis
    3. Non-enteric or unexplored fistulas
    4. Necrotic tissue with eschar remaining in the wound after surgical debridement (once necrotic tissue or eschar is removed from the wound bed, subjects may be included)
    5. Unprotected, exposed blood vessel, anastomotic sites, organs, or nerves in direct contact with foam
    6. Thoracic or abdominal cavities
    7. Unexplored wounds that may communicate with adjacent body cavities
13. Subject's targeted wound that is contraindicated with the control group device and not suitable for participating in the trial judged by investigator
14. Participation in another device or drug study within the past 30 days before screening or during study participation
15. Other subjects who are not suitable for participating in the trial judged by investigator.
16. Wounds that require more than 2 images in order to capture the entire wound. NOTE: each image must not exceed 20 cm in any one direction.
17. Wound presents on greater than 50% of the circumference of any part of the body (e.g. wound that wraps around >50% of a leg or arm).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhijun Pan, Director, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (4):
- China (4):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Foshan Hospital of TCM, Foshan, Guangdong
  - Xi'an Honghui Hospital, Xi’an, Shanxi
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Comparator Device: Negative Pressure Wound Drainage Material: A Negative pressure wound drainage material manufactured by Guangdong Shuangling Pharmaceutical Co., Ltd. (with unspecified pressures ranging from -150 to -380mmHg) was selected as the control group treatment device, which can apply the NPWT therapy with wall suction. This control device is widely used in clinical institutions in China to deliver NPWT. The target wound for each subject in both groups will be treated for up to 14 days or until deemed ready for closure by the investigator (whichever occurs first).
Period: Overall Study
Arm/Group | Investigational Device: V.A.C. VERAFLO™ Dressing Kit | Comparator Device: Negative Pressure Wound Drainage Material
Started | 84 | 86
Completed | 77 | 85
Not Completed | 7 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set. Among all 170 randomized subjects, 1 subject randomized to the investigational group was excluded from the full analysis set due to not receiving study NPWT after randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Device: V.A.C. VERAFLO™ Dressing Kit | Comparator Device: Negative Pressure Wound Drainage Material | Total
Number analyzed (Participants) | 83 | 86 | 169
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (10.97) | 47.5 (13.55) | 48.6 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 21 | 36
  Male | 68 | 65 | 133
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 83 | 86 | 169
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 83 | 86 | 169
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Definitive surgical debridement prior to enrollment [Count of Participants; unit: Participants]
  yes | 83 | 86 | 169
  no | 0 | 0 | 0
Baseline wound area (cm^2) [Mean (Standard Deviation); unit: cm^2] | 62.87 (50.402) | 50.16 (43.570) | 56.40 (47.340)
Baseline wound volume (cm^3) [Mean (Standard Deviation); unit: cm^3] | 20.31 (38.604) | 12.61 (16.264) | 16.41 (29.660)
Wound etiology/type [Count of Participants; unit: Participants]
  Traumatic | 55 | 68 | 123
  Surgical Dehisced | 22 | 15 | 37
  Pressure Ulcer | 0 | 0 | 0
  Diabetic Ulcer | 3 | 3 | 6
  other | 3 | 0 | 3
Wound age (days) [Mean (Standard Deviation); unit: days] | 24.44 (31.237) | 27.66 (29.798) | 26.08 (30.456)

OUTCOME MEASURES:

1. Primary Outcome: Wound Volume Reduction Rate (Unit: %)
Description: percent of total wound volume change relative to baseline over 14 days or until deemed ready for closure by investigator (whichever occurred first) over 14 days or until deemed ready for closure by investigator (whichever occurred first)
Time Frame: over 14 days or until deemed ready for closure by investigator (whichever occurred first)
Population: Per Protocol Set
Measure: Mean (Standard Deviation); unit: percentage of baseline wound volume
Arm/Group | Investigational Device: V.A.C. VERAFLO™ Dressing Kit | Comparator Device: Negative Pressure Wound Drainage Material
Number analyzed (Participants) | 60 | 61
percentage of baseline wound volume | 62.15 (43.485) | 65.04 (40.088)
Statistical Analysis 1: Comparison: Investigational Device: V.A.C. VERAFLO™ Dressing Kit vs Comparator Device: Negative Pressure Wound Drainage Material; Test type: Non-Inferiority — the non-inferiority margin is 20%; least square means difference = 0.89, 95% CI 2-sided [-14.30 to 16.07] — To establish non-inferiority the lower limit of the least square mean difference had to be > -20%

2. Secondary Outcome: Time to Completion of Wound Bed Preparation (Unit: Day)
Description: duration in days from the randomization until target wound ready for closure by secondary intervention judged by investigator.
Time Frame: Over 14 days or until deemed ready for closure by investigator (whichever occurred first)
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Investigational Device: V.A.C. VERAFLO™ Dressing Kit | Comparator Device: Negative Pressure Wound Drainage Material
Number analyzed (Participants) | 83 | 86
days | 9.0 [9.0 to 10.0] | 9.0 [9.0 to 10.0]

3. Secondary Outcome: Wound Area Reduction Rate (Unit: %)
Description: percent of total wound area change over 14 days or until deemed ready for closure by investigator (whichever occurred first)
Time Frame: Over 14 days or until deemed ready for closure by investigator (whichever occurred first)
Population: Per Protocol Set
Measure: Mean (Standard Deviation); unit: percentage of baseline wound area
Arm/Group | Investigational Device: V.A.C. VERAFLO™ Dressing Kit | Comparator Device: Negative Pressure Wound Drainage Material
Number analyzed (Participants) | 60 | 61
percentage of baseline wound area | 19.21 (23.267) | 27.20 (21.439)
Statistical Analysis 1: Comparison: Investigational Device: V.A.C. VERAFLO™ Dressing Kit vs Comparator Device: Negative Pressure Wound Drainage Material; Test type: Superiority; p = 0.24, ANCOVA; ANCOVA model had fixed effects of treatment arm, center and wound size

ADVERSE EVENTS:
Time Frame: up to 14 days
Arm/Group | Investigational Device: V.A.C. VERAFLO™ Dressing Kit | Comparator Device: Negative Pressure Wound Drainage Material
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/84 | 1/85
Other Adverse Events (participants affected / at risk) | 34/84 | 36/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Device: V.A.C. VERAFLO™ Dressing Kit (N=84) | Comparator Device: Negative Pressure Wound Drainage Material (N=85)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Investigational Device: V.A.C. VERAFLO™ Dressing Kit (N=84) | Comparator Device: Negative Pressure Wound Drainage Material (N=85)
Medical device site pain (General disorders) | 6 | 4
Pain (General disorders) | 4 | 6
Pyrexia (General disorders) | 1 | 3
Inflammation (General disorders) | 1 | 2
Hyperpyrexia (General disorders) | 1 | 0
Medical device site exfoliation (General disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 7 | 6
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 5 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Skin injury (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Blood pressure increased (Investigations) | 1 | 2
Blood glucose decreased (Investigations) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Hypercoagulation (Blood and lymphatic system disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-23): https://cdn.clinicaltrials.gov/large-docs/93/NCT05902793/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT05902793/SAP_001.pdf